CLINICAL TRIAL: NCT06292286
Title: Secondary Neoadjuvant Chemotherapy and Interval Cytoreductive Surgery in Platinum-sensitive Recurrent Epithelial Ovarian Cancer Patients - a Pilot Study
Brief Title: Secondary Interval Cytoreductive Surgery in Platinum-sensitive Recurrent Epithelial Ovarian Cancer
Acronym: SCENIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ka-Yu Tse, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 22-704
Record Dates: First submitted 2023-12-15; First posted 2024-03-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Cisplatin; Paclitaxel; Gemcitabine; liposomal doxorubicin; Bevacizumab; Biosimilar Pharmaceuticals; Cytoreduction Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Neoadjuvant carboplatin and paclitaxel followed by cytoreductive surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy and surgery arm (Experimental): Patients receive platinum-based chemotherapy with or without bevacizumab, and then undergo cytoreductive operation, for the first recurrence of EOC.
  Interventions: Procedure: Carboplatin or cisplatin; Drug: Paclitaxel, gemcitabine or liposomal doxorubicin with or without bevacizumab or biosimilar; Drug: Bevacizumab or biosimilar; Procedure: Cytoreductive surgery

INTERVENTIONS:
Procedure: Carboplatin or cisplatin — Carboplatin of cisplatin for 3-6 cycles
  Other Names: Paraplatin or Platinol
Drug: Paclitaxel, gemcitabine or liposomal doxorubicin with or without bevacizumab or biosimilar — Paclitaxel, gemcitabine or liposomal doxorubicin, for 3-6 cycles
  Other Names: Taxol, Gemzar, Caelyx
Drug: Bevacizumab or biosimilar — Optional
  Other Names: Avastin or mvasi
Procedure: Cytoreductive surgery — Cytoreductive surgery after chemotherapy

SUMMARY:
About 80% of advanced ovarian cancer patients recurred in 2-3 years. Secondary cytoreduction benefits selected patients who have high chance of complete resection. Whether secondary interval surgery can be used at recurrence is not known.

DETAILED DESCRIPTION:
Our study aims to evaluate the complete resection rate at interval cytoreductive surgery for recurrent ovarian cancer patients, and to determine the safety and survival outcomes of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed EOC, fallopian tube or primary peritoneal carcinoma
* >= 3 cycles of platinum-based chemotherapy, with or without bevacizumab and / or PARPi, at primary setting
* Platinum-free interval should be >=6 months from the last dose of platinum-based chemotherapy
* Upfront SCR not feasible
* Patients should have Eastern Cooperative Oncology Group (ECOG) performance score 0 to 2 within 28 days prior to recruitment.
* Patients must have adequate bone marrow, renal, hepatic and neurological function within 28 days prior to the start of treatment.

Exclusion Criteria:

* Non-epithelial or borderline tumors are excluded
* Patients who have with concurrent malignancy within five years (except for basal or squamous cell skin cancer, in-situ breast cancer, stage 1a grade 1-2 endometrioid endometrial carcinoma without lymphovascular invasion) are excluded.
* Patients using more than one line of chemotherapy are excluded.
* Patients who have platinum-resistant or refractory recurrence are excluded.
* Patients having second relapse or beyond are excluded.
* Patients who have contraindications to operation, e.g., unresolved thrombocytopenia, bowel obstruction in the last 4 weeks prior to enrolment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete resection rate | 12 months
  Rate of complete resection at the time of operation

SECONDARY OUTCOMES:
12-month progression-free survival rate | 12 months
  The time from the first dose of chemotherapy to the first documentation of objective tumor progression (PD) or to death due to any cause, whichever occurs first.
12-month overall survival rate | 12 months
  Overall survival is defined as the time from the first dose of chemotherapy to the date of death due to any cause.
Surgical complication rate | 12 months
  Complications are graded by the Clavien-Dindo classification
Quality of life scale | 12 months
  Different functional scales will be assessed by questionnaires like the EORTC questionnaires where all scales range from 0-100. The higher the score, the greater the intensity of that particular item is.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yu Tse, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong